CLINICAL TRIAL: NCT01399723
Title: Amoxicillin Versus Benzyl Penicillin for Severe Childhood Pneumonia Amongst Inpatients: An Open Label Randomised Controlled Non-inferiority Trial
Brief Title: Amoxicillin Versus Benzyl Penicillin for Treatment of Children Hospitalised With Severe Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KEMRI-Wellcome Trust Collaborative Research Program (Other)
Collaborators: University of Oxford (Other); London School of Hygiene and Tropical Medicine (Other); University of Nairobi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEMRI_CT_2010/0014; SSC 1911
Record Dates: First submitted 2011-07-12; First posted 2011-07-22 (Estimated); Results first posted 2015-02-13 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-01

CONDITIONS: Pneumonia
Keywords: Severe pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Amoxicillin; Penicillin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amoxicillin 45mg/kg 12 hourly (Experimental)
  Interventions: Drug: Amoxicillin
- Benzyl Penicillin 50,000IU/kg 6 hourly (Active Comparator)
  Interventions: Drug: Benzyl penicillin

INTERVENTIONS:
Drug: Amoxicillin — Oral 45mg/kg 12 hourly
  Arms: Amoxicillin 45mg/kg 12 hourly
Drug: Benzyl penicillin — Intravenous 50,000IU/kg 6 hourly
  Arms: Benzyl Penicillin 50,000IU/kg 6 hourly

SUMMARY:
This study seeks to determine whether clinical outcome following initial treatment of severe pneumonia with oral amoxicillin is as effective as the current standard benzyl penicillin. The study will also provide an estimate of the proportion of Kenyan children with severe pneumonia who fail treatment with a single antibiotic.

DETAILED DESCRIPTION:
Case management for the treatment of childhood acute respiratory infections has been widely promoted in many developing countries for over 20 years. Despite this, pneumonia continues to claim over 1.5 million lives of children under five annually. The use of affordable, easily-administered, safe, effective treatments can potentially reduce the burden of childhood pneumonia. The WHO recommends the use of a single antibiotic for the treatment of severe pneumonia. Whereas in Asia, evidence from large randomized clinical trials has changed policy recommendations for treatment of severe pneumonia from parenteral penicillin to oral amoxicillin, there is little evidence to inform a similar move in African children where pneumonia is associated with poorer outcomes. In this study the investigators will investigate effectiveness of oral amoxicillin versus the current standard treatment, benzyl penicillin in severe childhood pneumonia using a randomized controlled non-inferiority design preceded by a pilot pre-intervention phase. The investigators will also collect observational data HIV-exposed / infected children with severe pneumonia. 594 children aged 2 - 59 months admitted with clinical signs of severe pneumonia to up to 7 hospitals in Kenya will be randomly assigned to receive either oral amoxicillin or injectable benzyl penicillin. They will then be followed up for the primary outcome of pre-defined treatment failure at 48 hours. The results of this trial will provide valuable data on the effectiveness of oral amoxicillin in the treatment of severe pneumonia in a population of Kenyan children and determine the practicability of conducting large pragmatic trials on pneumonia in Africa similar to those done in Asia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs of WHO-defined severe pneumonia
* Age 2 months to 59 months

Exclusion Criteria:

* Clinical signs of WHO-defined very severe pneumonia
* Clinical or laboratory diagnosis of meningitis
* Clinical diagnosis of severe malnutrition (marasmus/kwashiorkor)
* Clinical or laboratory diagnosis of severe anaemia requiring transfusion
* HIV-exposure on rapid HIV antibody test (only observational data will be collected from these patients)
* Elimination of signs of severe pneumonia in a child with wheeze after outpatient bronchodilator therapy
* Chronic condition that may underlie or contribute to a presentation with respiratory distress such as: known chronic renal or cardiac disease, presence of cerebral palsy predisposing child to aspiration/hypostatic pneumonia
* Established bronchiectasis or congenital abnormality of the lower respiratory tract
* Upper airway obstruction producing stridor
* Admission from outpatient clinic specifically for treatment of TB
* Referral from another inpatient facility following treatment with injectable antibiotics for more than 24 hours or because the initial regimen is considered to have failed
* Documented history of >48hours treatment with oral amoxicillin
* Failure to obtain informed consent
* Penicillin allergy

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 561 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ambrose Agweyu, MSc, Principal Investigator — Kemri- Wellcome Trust Research Programme, Nairobi, Kenya; Elizabeth Obimbo, MMed, Principal Investigator — Department of Paediatrics and Child Health, University of Nairobi, Nairobi, Kenya; Roma Chilengi, MD, Principal Investigator — Centre for Infectious Disease Research, Zambia; Tansy Edwards, MSc, Principal Investigator — London School of Hygiene and Tropical Medicine; Mike English, MD, Principal Investigator — Kemri - Wellcome Trust Research Programme, Nairobi, Kenya
Locations (6):
- Kenya (6):
  - Kerugoya District Hospital, Kerugoya, Central
  - Embu Provincial General Hospital, Embu, Eastern
  - Mbagathi District Hospital, Nairobi, Nairobi County
  - Kisumu East District Hospital, Kisumu, Nyanza
  - New Nyanza Provincial General Hospital, Kisumu, Nyanza
  - Bungoma District Hospital, Bungoma, Western

REFERENCES:
- [Derived] Agweyu A, Gathara D, Oliwa J, Muinga N, Edwards T, Allen E, Maleche-Obimbo E, English M; Severe Pneumonia Study Group. Oral amoxicillin versus benzyl penicillin for severe pneumonia among kenyan children: a pragmatic randomized controlled noninferiority trial. Clin Infect Dis. 2015 Apr 15;60(8):1216-24. doi: 10.1093/cid/ciu1166. Epub 2014 Dec 30. PMID 25550349

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amoxicillin 45mg/kg 12 Hourly | Benzyl Penicillin 50,000IU/kg 6 Hourly
Started | 263 | 264
Completed | 263 | 263
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Amoxicillin: Amoxicillin 45mg/kg 12 hourly
- Penicillin: Benzyl penicillin 50000 IU 6 hourly
- Total: Total of all reporting groups
Arm/Group | Amoxicillin | Penicillin | Total
Number analyzed (Participants) | 263 | 264 | 527
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14 [7 to 25] | 13 [7 to 24] | 13 [7 to 24]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 106 | 226
  Male | 143 | 158 | 301
Region of Enrollment [Number; unit: participants]
  Kenya | 263 | 264 | 527

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure at 48 Hours (Two Full Days After Enrollment)
Description: Development of any signs of very severe pneumonia at any time Hypoxemia defined as SpO2 <85% or <80% for altitude < or ≥1500m respectively measured after minimum of 3 minutes on ambient air Persistent vomiting (occurring within 30 minutes of administration of amoxicillin with failure to retain drug after 3 successive attempts at administration) at any time Clinical diagnosis of new bacterial co-morbid condition requiring revision of antibiotic treatment at any time Lower chest wall indrawing Temperature ≥38◦C Respiratory rate ≥5bpm of admission rate if above age-adjusted normal upper limit
Time Frame: 48 hours
Population: Intention to treat analysis
Measure: Number; unit: participants
Groups:
- Penicillin: Benzyl penicillin 50000 IU/kg 6 hourly
Arm/Group | Amoxicillin | Penicillin
Number analyzed (Participants) | 263 | 263
participants | 20 | 21
Statistical Analysis 1: Comparison: Amoxicillin vs Penicillin; Test type: Non-Inferiority or Equivalence — Noninferiority between amoxicillin and benzyl penicillin was defined a priori as a risk difference of treatment failure and associated upper bound of the 95% confidence interval (CI) of <7%. A sample size of 576 would provide 80% power to detect noninferiority of amoxicillin against benzyl penicillin within a margin of 7% at a 1-sided level of significance of 0.025, assuming a prevalence of treatment failure of 10% at 48 hours derived from a preintervention pilot phase of the study; Risk Difference (RD) = -0.4, 95% CI 2-sided [-5.0 to 4.2] — Risk difference comparison is for amoxicillin versus benzyl penicillin

2. Secondary Outcome: Treatment Failure at or Before Discharge / Day 5 Post Enrollment (Whichever Occurs First)
Description: Treatment failure as defined in the primary outcome measure.
Time Frame: Patients will be followed up from the day of hospitalisation (day 0) until the day of medical discharge (average duration of 3 days) or until day 5 of hospitalisation (whichever occurs first).
Population: Intention to treat analysis
Measure: Number; unit: participants
Groups:
- Penicillin: Benzyl Penicillin 50,000IU/kg 6 hourly
Arm/Group | Amoxicillin | Penicillin
Number analyzed (Participants) | 263 | 263
participants | 30 | 29
Statistical Analysis 1: Comparison: Amoxicillin vs Penicillin; Test type: Non-Inferiority or Equivalence — The initial sample size estimate of 576 children (288 per group) would provide 80% power to detect noninferiority of amoxicillin against benzyl penicillin within a margin of 7% at a 1-sided level of significance of 0.025, assuming a prevalence of treatment failure of 10% at 48 hours derived from a preintervention pilot phase of the study; Risk Difference (RD) = 0.4, 95% CI 2-sided [-5.0 to 5.8] — Risk difference comparison is for amoxicillin versus benzyl penicillin

3. Secondary Outcome: Readmission With Diagnosis of Severe or Very Severe Pneumonia Within 14 Days of Enrollment
Time Frame: Day 0 to Day 14
Reporting Status: Not Posted

4. Secondary Outcome: Death at or Before Five Days Following Enrollment
Description: Death defined as: in-hospital death occurring at any time after randomisation (recruitment for HIV-exposed participants) or verbal report of death of the enrolled patient from parent/guardian communicated either directly or via telephone conversation.
Time Frame: Day 0 to Day 5
Reporting Status: Not Posted

5. Secondary Outcome: Outcome (Death/Readmission) at 14 Days as Determined by Telephone or Direct Interview
Description: Definition of death as described in third secondary outcome measure.
Time Frame: Day 14
Measure: Number; unit: participants
Arm/Group | Amoxicillin | Penicillin
Number analyzed (Participants) | 244 | 250
participants | 33 | 42
Statistical Analysis 1: Comparison: Amoxicillin vs Penicillin; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Risk Difference (RD) = -3.3, 95% CI 2-sided [-10.0 to 3.0] — Risk difference comparison is for amoxicillin versus benzyl penicillin

ADVERSE EVENTS:
Groups:
- Benzyl Penicillin: Benzyl Penicillin 50,000IU/kg 6 hourly
Arm/Group | Amoxicillin | Benzyl Penicillin
Serious Adverse Events (participants affected / at risk) | 1/263 | 3/263
Other Adverse Events (participants affected / at risk) | 0/263 | 0/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amoxicillin (N=263) | Benzyl Penicillin (N=263)
Congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Hypovolemic shock (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) — Acute on chronic kidney disease
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No